CLINICAL TRIAL: NCT03397836
Title: Health TAPESTRY Ontario: A Randomized Controlled Trial
Brief Title: Health TAPESTRY Ontario
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Red Cross (Other); Ontario Ministry of Health and Long Term Care (Other Government); David Braley (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3967
Record Dates: First submitted 2017-12-12; First posted 2018-01-12 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2020-11

CONDITIONS: Aging
Keywords: Older adults; Optimal aging; Primary health care; Randomized control trial; Integrated care; Health care volunteers; interdisciplinary health care teams; Implementation; Health services research; Patient centered care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health TAPESTRY Intervention (Experimental): This patient group will begin receiving the TAPESTRY interventions from time zero
  Interventions: Other: Health TAPESTRY Intervention
- Usual Care (Active Comparator): This patient group will receive the intervention after a 6 month waiting period. In the first 6 months they will receive usual care and they will be used as a comparison group.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Health TAPESTRY Intervention — The patient will receive in-home visits from trained volunteers who will collect information electronically using a tablet computer. The volunteers will collect information about the client's health goals, health risks, and needs using a specifically designed application (TAP-App). Once the data is gathered, it is summarized into a report (TAP-report) which is securely and electronically sent to the health care clinic (TAP huddle). The team can leverage clinic supports and/or community supports as they deem appropriate to help clients reach their health goals and address any needs and risks which were reported during the volunteer visits.
  Arms: Health TAPESTRY Intervention
Other: Usual Care — Usual care while waiting for the Health TAPESTRY intervention, the control group will receive usual care from their healthcare providers.
  Arms: Usual Care

SUMMARY:
The Health Teams Advancing Patient Experience: Strengthening Quality (Health TAPESTRY) is a community-based program led by primary care teams, that creates connections between trained community volunteers, interprofessional health care teams, novel technology and community engagement through improved system navigation. The overall vision is to help people stay healthier for longer in the places where they live.

DETAILED DESCRIPTION:
The Health Teams Advancing Patient Experience: Strengthening Quality (Health TAPESTRY) involves recording a person's life and health goals, screening for health risks and needs, and then initiating a plan that supports achievement of those goals and address risks and needs. It includes four parts:

1. Trained volunteers connect with clients (patients) in their home to gather health and social information and discuss and record life and health goals
2. Interprofessional health care teams provide health care services to the client and focuses on a plan to support them on meeting their health goals
3. Technology is used to collect and share information
4. Community engagement connects clients with resources and supports in the community

Initial findings from Implementation Phase I: 6-month unblinded delayed intervention pragmatic randomized controlled trial that took place in Hamilton, ON (HiREB File #14-726, Clinical Trials.gov NCT02283723) showed significant differences between the intervention and control group. Specifically, at 6-months the it was found:

* a reduction in the intervention group versus control group in self-reported time sitting
* an increase in minutes walking in the intervention group versus the control group
* an increase in number of primary care visits in the intervention group versus the control group
* a reduction in odds of people experiencing 1 or more hospitalizations in the intervention group versus the control group

Understanding the feasibility of implementing Health TAPESTRY in other primary care sites is important to evaluate its potential as an approach. Replication of these initial findings are critical in terms of empirical support for the approach as well as spread and scalability in the wider primary health care system.

Six sites have been identified as Health TAPESTRY-Ontario implementation sites. It should be noted that all appropriate site approvals will be obtained prior to implementation.

1. Niagara North Family Health Team (Niagara-on-the-Lake) (Mary Keith, executive Lead; Dr. Karen Berti, family health team lead)
2. McMaster Family Health Team (Hamilton) (Doug Oliver, family health team lead)
3. Superior Family Health Team (Sault Ste Marie) (Michelle Brisbois, executive lead, Dr. Sarah White, family health team lead)
4. Dufferin and Area Family Health Team (Dufferin County) (Lianne Barbour, executive Lead, Dr. Mercedes Rodriguez, family health team lead)
5. Windsor Family Health Team (Windsor and surrounding area) (Sara Dalo, executive lead)
6. Harrow Family Health Team (Harrow and surrounding communities) (Margo Reilly, executive lead, Dr. Alexandra Lindberg, family health team lead)

A broad alliance between Canadian Red Cross and the Department of Family Medicine has been made, with Health TAPESTRY being a part of that alliance. As part of this partnership, the Canadian Red Cross partner will recruit, train, schedule, and retain community volunteers to operate in the 6 sites.

ELIGIBILITY:
Participant Inclusion Criteria:

* Be 70 years of age or older
* Rostered to a participating family physician

Participant Exclusion Criteria:

* They are expected to die within 12 months
* They live in a long-term care facility
* They (or their caregiver) are unable to speak and understand English
* They have other conditions or circumstances that means the patient is unable to engage with the volunteers or complete the TAP-App (e.g., severe dementia)
* They are out of the country for more than 6 months or otherwise unavailable for the intervention and assessments
* Participated in Health TAPESTRY phase I implementation (for Hamilton site)

Site Inclusion Criteria:

A Health TAPESTRY site must have the commitment and capacity to implement and sustain the full Health TAPESTRY Program (all four parts). As such, the following success factors are essential:

* A strong Lead Organization with a clearly identified Health TAPESTRY Practice Model Champion from primary care;
* Visible and influential primary care partner in governance and implementation;
* Team-based use of an electronic system for documentation;
* Primary care team available to provide core of implementation;
* Available Information Technology capacity and commitment to integrate with TAP-App (minimum HL7 document transfer capability) and kindred PHR within 6-9 months of program start date;
* Volunteer infrastructure that can recruit, train, sustain, and coordinate/schedule volunteers, and ensure volunteers have access to the digital health tools needed to fulfill role;
* Existing partnerships with local community services;
* Capacity for local program management either through existing staff or with the addition of new staff;
* Available in-kind resources that can support participation in the Health TAPESTRY Program (e.g., clinician and staff engagement, community engagement, patient engagement, etc.); and
* Commitment to evaluation including, but not limited to, collecting and sharing data from electronic documentation system (based on consent).

Site Exclusion Criteria:

* No functional primary care team linkage to support individual patient or client assessments
* Focused assessment on a single condition or disease

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 599 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
Change in Hospitalizations | Change of number of hospitalizations from baseline to 6 months
  Number of hospitalizations in the past 6 months.
Change in Physical activity | Change in physical activity from baseline measurement to 6 months
  Physical activity will be measured by the Short version of the International Physical Activity Questionnaire. Respondents indicate how many days in the past seven days and for how many minutes they have engaged in vigorous and moderate intensity activity and walking activity. Scores are calculated by multiplying the days by the number of minutes on one day, by the metabolic equivalent of task (8.0,4.0 and 3.3 for vigorous, moderate, walking activity respectively). Minimum score is of the scale is zero, with higher scores representing higher levels of physical activity.

SECONDARY OUTCOMES:
Emergency department and urgent care visits | Baseline, 6 months
  Number of emergency department and urgent care visits in the past 6 months. Reasons for each visit will also be extracted in order to describe the nature of visits.
Falls | Baseline, 6 months
  Number of falls in the past 6 months (those resulting in medical treatment).
Hours sitting | Baseline, 6 months
  Hours sitting will be measured by the sitting item on the Short version of the International Physical Activity Questionnaire. Respondents indicate for how many hours they sit in a typical day. Scale ranges from 0 hours to 24 hours, higher scores indicate higher hours sitting.
Patient enablement | Baseline, 6 months
  A modified version of the Patient Enablement Instrument will be used as a measure of patient empowerment in their own care. Specifically, the stem "as a result of your visit to the doctor today…" was deleted and instead, "after a usual visit with your family health care team, do you feel that you are…" was used.
Quality of life | Baseline, 6 months
  The EuroQol five dimension (EQ-5D-5L) will be used to measure quality of life. This survey asks respondents to rate their ability in five different domains: mobility, self-care, usual activities, pain, and anxiety/depression. In addition, respondents are asked to rate their current health state on a scale from 0 ('worst health you can imagine') to 100 ('best health you can imagine'). A score from the five domains is calculated using a macro program and ranges from 0 to 1.
Treatment burden | Baseline, 6 months
  Treatment burden will be measured by the Brief Treatment Burden Scale. Respondents are asked to rate their level of difficulty they have with ten different treatment-related tasks on a scale from "not difficult" to "extremely difficult".
Disease burden | Baseline, 6 months
  Disease burden will be measured using the Disease Burden survey. Respondents are asked to indicate which conditions they have, and for those conditions present, the degree to which the condition hurts their daily activity from "not at all" to "a lot". The list contains common chronic conditions.
Medications | Baseline, 6 months
  Number of long-term prescription medications (defined as use of a medication for 3 or more months).
Negative effects (unmet expectations) | Baseline, 6 months
  A measure of unmet expectations specifically developed for this trial. Participants will be asked to rate the level of their expectation with the question: 'In thinking about the kind and amount of care you received as a result of Health TAPESTRY, to what extent did it meet your expectations?' Answer option include: exceeded expectations, met expectations, no real difference in kind or amount of care received, or kind and amount of care received was worse than before Health TAPESTRY.
Negative effects (effects of labeling) | 6 months
  The negative effects of labeling will be measured using a survey developed for this trial. For those identifying that Health TAPESTRY made them aware of health conditions or risks they were unaware of before, an open-ended question to describe the impact of this awareness will be asked.
Negative effects (serious adverse events) | 6 months
  Serious adverse events will be recorded using retrospective chart audit.
Primary care visits | Baseline, 6 months
  Number of primary care visits.
Reason for hospitalization | Baseline, 6 months
  Reason for each hospitalization will be categorized into ambulatory care sensitive conditions or acute care conditions.

OTHER OUTCOMES:
Best and worst parts of intervention | 12 months
  Open-ended list of the five best and five worst parts of Health TAPESTRY for patients and health care providers.
Recommend to others | 6-months post intervention (patients), 12-months (healthcare providers)
  Patients and health care providers asked whether or not they would recommend Health TAPESTRY to others.
Satisfaction with volunteer | 6 months
  Satisfaction with interpersonal relationships with volunteer survey completed by patients.
Type of primary care visit | 6 months
  Recorded profession of the clinician holding the visit with the patient.
Length of hospital stay | 6 months
  Number of days spent in the hospital. Same-day hospitalizations will reflect zero days spent in the hospital for that particular hospitalization.
Critical incidents | 12 months
  Number and type of critical incidents will be tracked electronically.
Implementation processes | 1 months, 2 months, 3 months, 6 months, 9 months, 12 months
  NoMAD survey

CONTACTS AND LOCATIONS:
Overall Officials: Dee Mangin, MBChB,DPH,FR, Principal Investigator — McMaster University
Locations (1):
- Department of Family Medicine, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mangin D, Lamarche L, Oliver D, Blackhouse G, Bomze S, Borhan S, Carr T, Clark R, Datta J, Dolovich L, Gaber J, Forsyth P, Howard M, Marentette-Brown S, Risdon C, Talat S, Tarride JE, Thabane L, Valaitis R, Price D. Health TAPESTRY Ontario: A Multi-Site Randomized Controlled Trial Testing Implementation and Reproducibility. Ann Fam Med. 2023 Mar-Apr;21(2):132-142. doi: 10.1370/afm.2944. PMID 36973055
- [Derived] Lamarche L, Clark RE, Parascandalo F, Mangin D. The implementation and validation of the NoMAD during a complex primary care intervention. BMC Med Res Methodol. 2022 Jun 19;22(1):175. doi: 10.1186/s12874-022-01655-0. PMID 35718763
- [Derived] Gaber J, Datta J, Clark R, Lamarche L, Parascandalo F, Di Pelino S, Forsyth P, Oliver D, Mangin D, Price D. Understanding how context and culture in six communities can shape implementation of a complex intervention: a comparative case study. BMC Health Serv Res. 2022 Feb 17;22(1):221. doi: 10.1186/s12913-022-07615-0. PMID 35177040
- [Derived] Mangin D, Lamarche L, Oliver D, Bomze S, Borhan S, Browne T, Carr T, Datta J, Dolovich L, Howard M, Marentette-Brown S, Risdon C, Talat S, Tarride JE, Thabane L, Valaitis R, Price D. Health TAPESTRY Ontario: protocol for a randomized controlled trial to test reproducibility and implementation. Trials. 2020 Aug 14;21(1):714. doi: 10.1186/s13063-020-04600-y. PMID 32795381
- See also: Health TAPESTRY website — http://healthtapestry.ca/